CLINICAL TRIAL: NCT07050212
Title: A Comparative Study of the Application of Remimazolam, Dexmedetomidine, and Esketamine in Pediatric Preoperative Sedation
Brief Title: Application of Remimazolam, Dexmedetomidine, and Esketamine in Pediatric Preoperative Sedation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MCHH_013
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Remimazolam; Dexmedetomidine; Esketamine
MeSH Terms: interventions — remimazolam; Dexmedetomidine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam group: Remimazolam is administered intravenously at a dose of 0.3 mg/kg (Experimental): Remimazolam is administered intravenously at a dose of 0.3 mg/kg
  Interventions: Drug: remimazolam group
- dexmedetomidine group: dexmedetomidine is administered intravenously at a dose of 1 μg/kg (Active Comparator): dexmedetomidine is administered intravenously at a dose of 1 μg/kg
  Interventions: Drug: dexmedetomidine group
- esketamine group: esketamine is administered intravenously at a dose of 0.5 mg/kg (Active Comparator): esketamine is administered intravenously at a dose of 0.5 mg/kg
  Interventions: Drug: esketamine group

INTERVENTIONS:
Drug: remimazolam group — remimazolam is administered intravenously at a dose of 0.3 mg/kg
  Other Names: remimazolam
  Arms: Remimazolam group: Remimazolam is administered intravenously at a dose of 0.3 mg/kg
Drug: dexmedetomidine group — dexmedetomidine is administered intravenously at a dose of 1 μg/kg
  Other Names: dexmedetomidine
  Arms: dexmedetomidine group: dexmedetomidine is administered intravenously at a dose of 1 μg/kg
Drug: esketamine group — esketamine is administered intravenously at a dose of 0.5 mg/kg
  Other Names: esketamine
  Arms: esketamine group: esketamine is administered intravenously at a dose of 0.5 mg/kg

SUMMARY:
By comparing the application effects of three drugs in pediatric preoperative sedation, this study explores the optimal medication regimen, aiming to provide safer, more effective, and more personalized medication options for pediatric preoperative sedation. Additionally, this research will also focus on the impact of these three drugs on postoperative agitation in children, offering valuable references for the overall management of pediatric surgical anesthesia.

DETAILED DESCRIPTION:
Participants will be randomly allocated to three groups: remimazolam group(Group A), dexmedetomidine group(Group B), esketamine group(Group C). Before entering the operating room, an intravenous access is established. Under the accompaniment of a parent, one of the three drugs is administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 2 to 5 years old
2. the American Society of Anesthesiologists (ASA) physical status of Class I
3. scheduled for adenotonsillectomy under general anesthesia, will be included.

Exclusion Criteria:

1. Abnormal lung function and respiratory system function
2. airway obstruction or deformity, history of mental illness
3. electrocardiogram indicating bradycardia
4. history of cardiac disease

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Sedation success rate | 0, 3, 5, 10 minutes after the drug injection
  1 points represents the child being restless and irritable; 2 points represents that the child is quiet and cooperative; 3 points represents that the child is drowsy and able to obey instructions; A score of 4 indicates that the child is in a shallow sleep state and can be quickly awakened; 5 points represent the child falling asleep and having a slow response to calls; 6 points represent the child's deep sleep state and no response to calls. If the Ramasay score greater than 2 points, it is considered a successful sedation.
Onset time of sedation | 0, 3, 5, 10 minutes after the drug injection
  The time from the end of drug injection until the Ramsay score is greater than 2 points. If the Ramasay score greater than 2 points, it is considered a successful sedation. 1 points of ramasay scorere presents the child being restless and irritable; 2 points represents that the child is quiet and cooperative; 3 points represents that the child is drowsy and able to obey instructions; A score of 4 indicates that the child is in a shallow sleep state and can be quickly awakened; 5 points represent the child falling asleep and having a slow response to calls; 6 points represent the child's deep sleep state and no response to calls.
Parent-Child Separation Anxiety Score (PASA Score) | 0, 3, 5, 10 minute after the drug injection
  if the PASA score is greater than 2, it is considered a positive reaction to separation anxiety. 1 point represents that the child is easily separated from their parents；A score of 2 indicates that the child has crying sounds, easily comforted, and does not rely on their parents；A score of 3 indicates that the child is crying and cannot be comforted, but does not rely on their parents；4 points represent the child crying and relying on their parents

SECONDARY OUTCOMES:
Mask Acceptance Score (MAS) | 0, 3, 5, 10 minutes after the drug injection
  The MAS scale is used to evaluate the acceptance of respiratory masks in pediatric patients. Less than 2 points indicate satisfactory acceptance. 1 point represents that the child is fearless and easily accepts face masks; 2 points represent that the child is mildly fear of the face mask and easily be comfort; 3 points represent that the child is moderatly fear of the face mask and cannot be comforted; 4 points represent that the child is very afraid of the face mask and crying
incidence of adverse reactions | during intravenous bolus administration of sedative drugs and anesthesia induction
restlessness rating scale for awakening period(PAED) | 0, 5, 10, 20 minutes after the patient awake
  When the PAED score is greater than 2 points, the child is identified as agitated during the recovery period; if the PAED score is greater than 10 points, the child is identified as delirium in the awakening period.
Heart rate | 0, 3, 5, and 10 minutes after the drug injection
blood pressure | 0,3,5,10 minute after drug injectuion
  systolic pressure and diastolic pressure
respiratory rate | 0,3,5,10 minute after drug injectuion
pulse oximetry saturation | 0,3,5,10 minute after drug injectuion

CONTACTS AND LOCATIONS:
Overall Officials: Na Li NaLi, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
I plan to share IPD after the end of this study, including the study protocol, informed consent form and clinical study report.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: after the end of this study
Access Criteria: all